CLINICAL TRIAL: NCT06233643
Title: The Efficiency of Acupuncture Combined Intradermal Sterile Water Application in Acute Renal Colic: a Randomised Clinical Trial.
Brief Title: The Efficiency of Acupuncture Combined Intradermal Sterile Water Application in Acute Renal Colic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Third Affiliated Hospital of Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Jianghua Yang, Urologist of Third BUCM,MD, The Third Affiliated Hospital of Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ThirdBUCM
Record Dates: First submitted 2024-01-13; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Renal Colic
Keywords: Acupuncture; Intradermal Sterile Water; NSAIDS
MeSH Terms: conditions — Renal Colic | interventions — Phloroglucinol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group received acupuncture combined with intradermal sterile water (Experimental): These acute renal colic patients who will received acupuncture combined with intradermal sterile water
  Interventions: Combination Product: Acupuncture Combined Intradermal Sterile Water
- The group received intramuscular inject phloroglucinol (Active Comparator): These acute renal colic patients who will received intramuscular inject phloroglucinol.
  Interventions: Drug: Phloroglucinol

INTERVENTIONS:
Drug: Phloroglucinol — The active comparators will be treated with 40 mg of Phloroglucinol in the form of a single intramuscular injection.
  Arms: The group received intramuscular inject phloroglucinol
Combination Product: Acupuncture Combined Intradermal Sterile Water — Acupuncture was applied to a seated patient using the urinary bladder meridian points and combianed Intradermal Sterile Water in costovertebral area where the patient's pain was located (Sterile water of 0.5 ml was injected as intradermal into 4 points at a depth of 1-3 mm to form papules)
  Arms: The group received acupuncture combined with intradermal sterile water

SUMMARY:
The goal of this clinical trial is to compare the analgesic effect and tolerance profile of acupuncture combined with intradermal sterile water application versus intramuscular phloroglucinol in acute renal colic. In this study, we aimed primarily to test the efficacy of acupuncture combined with intradermal sterile water application as a rapid and effective treatment in severe renal colic.

Participants will randomly divided into two groups. The first group received only intramuscular phloroglucinol, the second group received acupuncture and intradermal sterile water.The visual analog scale (VAS,ranging from 0 for no pain to 10 for maximum imaginable pain) was used to assess pain intensity at baseline and at 10, 20, 30, 45,and 60 minutes following the start of the treatment protocol. Possible treatment side effects were also recorded.

DETAILED DESCRIPTION:
Inclusion criteria：We included all consecutive patients aged >18 years and presenting to our medical center with uncomplicated acute renal colic. Renal colic was considered if the patient description of pain included sudden onset of symptoms; unilateral flank or lower abdomen pain; irradiation to the back, side, or groin region; urination problems, including urinating difficultly and/or an abnormally dark or red urine; and the absence of other obvious conditions explaining patient symptoms.

Exclusion criteria:We excluded patients with complicated acute renal colic, defined by the presence of bilateral pain, fever, and/or decreased urine output (<500 mL per day). Patients presenting with posttraumatic pain, those taking anticoagulant medications or with coagulation problems, those with skin afflictions (infections, hematoma, dermatosis) that would impair the use of certain acupuncture points, those unable to assess the degree of pain using the VAS, those who had received analgesics in the 6 hours prior to enrollment, those refusing or unable to give written consent, and pregnant women were also excluded from this study. All participants read and signed the informed consent form of the study, which was approved by the ethics committee of the Third Affiliated Hospital of Beijing University of Chinese Medicine.

ELIGIBILITY:
Inclusion criteria：We included all consecutive patients aged >18 years and presenting to our medical center with uncomplicated acute renal colic. Renal colic was considered if the patient description of pain included sudden onset of symptoms; unilateral flank or lower abdomen pain; irradiation to the back, side, or groin region; urination problems, including urinating difficultly and/or an abnormally dark or red urine; and the absence of other obvious conditions explaining patient symptoms.

Exclusion criteria:We excluded patients with complicated acute renal colic, defined by the presence of bilateral pain, fever, and/or decreased urine output (<500 mL per day). Patients presenting with posttraumatic pain, those taking anticoagulant medications or with coagulation problems, those with skin afflictions (infections, hematoma, dermatosis) that would impair the use of certain acupuncture points, those unable to assess the degree of pain using the VAS, those who had received analgesics in the 6 hours prior to enrollment, those refusing or unable to give written consent, and pregnant women were also excluded from this study. All participants read and signed the informed consent form of the study, which was approved by the ethics committee of the Third Affiliated Hospital of Beijing University of Chinese Medicine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Baseline characteristics of patients | before treatment
  Baseline characteristics of patients between two groups concerning age (years), sex (male or female ）, and baseline VAS score (ranging from 0 for no pain to 10 for maximum imaginable pain)
primary outcome | 10, 30, 60, and 120 minutes after treatment.
  Visual analogue scale (VAS, ranging from 0 for no pain to 10 for maximum imaginable pain) will be used to assess pain intensity after 10, 30, 60, and 120 minutes.

SECONDARY OUTCOMES:
side effects | in 120 minutes after treatment.
  Document any side effects that occur after the intervention